CLINICAL TRIAL: NCT00773409
Title: A Prospective Study Evaluating the Incidence of Nephrogenic Systemic Fibrosis in Patients With Stages 4 to 5 Chronic Kidney Disease Without Exposure to Gadolinium Based Contrast Agents Within the Past 10 Years
Brief Title: Evaluation of the Risk of Nephrogenic Systemic Fibrosis (NSF) in Patients With Chronic Kidney Disease Without Exposure to Gadolinium Based Contrast Agents (GBCA)
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: NSF-101
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed tissue samples and tissue sample for testing of GBCA.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this long term study is to prospectively evaluate the incidence of NSF in patients with severe CKD or kidney failure including patients undergoing dialysis (stages 4 and 5 i.e., with an eGFR below 30)who have not had exposure to a GBCA within 10 years prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Has CKD with an eGFR below 30 mL/min/1.73m2 and/or undergoing dialysis as calculated from a serum creatinine (SCr) value obtained from the local laboratory within 24 hours prior to signing the informed consent;
* Provides written informed consent and is willing to comply with protocol requirements

Exclusion Criteria:

* Has received a GBCA within the past 10 years prior to inclusion in this study including the administration of a GBCA for something other than an MRI (e.g., CT or DSA);
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data and achieving study objectives;
* Has ever been suspected of, or diagnosed with, NSF;
* Is unable or unwilling to return for necessary office visits, to be examined by dermatologists or to undergo deep skin biopsy and laboratory/other diagnostic evaluations should development of NSF be suspected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 400 patients will be enrolled into this study based on their renal function (eGFR) and the fact that they have been GBCA free for the past 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence of NSF in patients that have not been exposed to GBCA within the last 10 years with severe CKD including those undergoing dialysis observed during the follow-up time period over the total number of eligible patients. | 1,3,6,12,18,24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics Inc., Princeton, New Jersey, United States